CLINICAL TRIAL: NCT02499614
Title: Crizotinib in Pretreated Metastatic Non-small-cell Lung Cancer With MET Amplification or MET Exon 14 Mutation or ROS1 Translocation (METROS)
Brief Title: Crizotinib in Pretreated Metastatic Non-small-cell Lung Cancer With MET Amplification or ROS1 Translocation (METROS)
Acronym: METROS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoRT 01/2014
Record Dates: First submitted 2015-03-30; First posted 2015-07-16 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: MET amplification; ROS1 translocation; Crizotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with MET amplification or MET exon 14 mutation (Experimental): Pretreated NSCLC patients with MET amplification or MET exon 14 mutation with locally advanced or metastatic NSCLC and with at least one measurable tumor lesion will be considered eligible for the trial and they will receive crizotinib 250 mg BID p.o until disease progression, unacceptable toxicity or patient refusal.
  Interventions: Drug: Crizotinib
- Patients with ROS1 translocation (Experimental): Pretreated NSCLC patients with ROS1 translocation with locally advanced or metastatic NSCLC and with at least one measurable tumor lesion will be considered eligible for the trial and they will receive crizotinib 250 mg BID p.o until disease progression, unacceptable toxicity or patient refusal.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Eligible patients with ROS1 translocation or MET amplification will be treated with Crizotinib at the standard dose of 250 mg BID. The dose of crizotinib may be adjusted depending on the type and severity of toxicity encountered
  Other Names: XALKORI

SUMMARY:
Phase II, two arms, parallel, non comparative study with crizotinib in patients with ROS 1 translocation or MET amplification or MET exon 14 mutation

DETAILED DESCRIPTION:
This is a phase II, prospective, two arms, parallel, non comparative study with crizotinib in pretreated NSCLC patients with ROS1 translocation or MET amplification or MET exon 14 mutation (figure 1). Patients with locally advanced or metastatic NSCLC, pretreated with at least one previous chemotherapy line and with at least one measurable tumor lesion will be considered eligible for the trial. All potentially eligible patients will be evaluated for MET and ROS1 by FISH to detect MET amplification or ROS1 translocation. MET mutation will be assessed using direct sequencing or high sensitive methods. After evaluation of inclusion and exclusion criteria, and after signature of informed consent form, all MET amplified or MET exon 14 mutation or ROS1 translocated eligible patients will receive crizotinib 250 mg BID p.o until disease progression, unacceptable toxicity or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of NSCLC
* Availability of tumor tissue for ROS1 and MET analyses
* Patient positive for ROS1 translocation or MET amplification
* At least one radiological measurable disease according to RECIST criteria (Response Evaluation Criteria in Solid Tumors )
* At least 1 previous standard chemotherapy regimen
* Performance status 0-2 (ECOG)
* Patient compliance to trial procedures
* age ≥ 18 years
* Written informed consent
* Adequate BM function (ANC ≥ 1.5x109/L, Platelets ≥ 100x109/L, HgB > 9g/dl)
* Adequate liver function (bilirubin <G2, transaminases no more than 3xULN/<5xULN in present of liver metastases).
* Normal level of alkaline phosphatase and creatinine.
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of approved contraceptive method [intrauterine contraceptive device (IUD), birth control pills, or barrier device] during and for ninety(90) days after end of treatment.

Exclusion Criteria:

* No tumor tissue available or patient negative for ROS1 translocation or MET amplification
* Absence of any measurable lesion
* For ROS1+ patients: Previous therapy with crizotinib or any anti-ALK agent
* For MET amplified patients: Evidence of MET amplification in tumor tissue collected in EGFR mutant patient at time of EGFR-TKI acquired resistance occurrence. An EGFR mutant patient is eligible if MET amplification is detected in a tumor specimen collected before starting an EGFR-TKI
* No previous chemotherapy
* Concomitant radiotherapy or chemotherapy.
* Previous radiotherapy on the target lesion(s). If all sites were included in radiotherapy fields patient is eligible only if there is evidence of progressive disease after completion of radiotherapy.
* Symptomatic brain metastases
* Diagnosis of any other malignancy during the last 5 years, except for in situ carcinoma of cervix uteri and squamous cell carcinoma of the skin
* Pregnancy or lactating
* Other serious illness or medical condition potentially interfering with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Response rate to crizotinib in patients with ROS1 translocation or MET amplification or MET exon 14 mutation | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months
Overall Survival (OS) | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months
Toxicity analysis: Incidence of Grade 3-4 Grade Toxicity graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0 | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months
Correlation with additional tumor biomarkers in tumor tissue or blood | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months
Response according to different levels of ROS1 translocation or MET amplification (ratio >2.2 and <5 versus ratio ≥ 5) or MET exon 14 mutation | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Crinò, Principal Investigator — Ospedale Santa Maria della Misericordia - Azienda Ospedaliera di Perugia
Locations (26):
- Italy (26):
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)- Oncologia Medica, Meldola, Forlì- Cesena
  - Ospedale Versilia- Oncologia, Camaiore, Lucca
  - Ospedale per gli Infermi - Presidio Ospedaliero di Faenza- Unità Operativa di Oncologia Medica, Faenza, Ravenna
  - Ospedale Umberto I°- Unità Operativa di Oncologia, Lugo, Ravenna
  - A. O. "Ospedale di Circolo" di Busto Arsizio- Struttura Complessa di Oncologia Medica, Saronno, Varese
  - Sacro Cuore- Don Calabria Hospital- U.O.C. Oncologia Medica, Negrar, Verona
  - Istituto Toscano Tumori Ospedale San Donato- U.O.C. di Oncologia Medica Dipartimento di Oncologia USL-8, Arezzo
  - Azienda Ospedaliera di Rilievo Nazionale "S.G. Moscati"- U.O. di Oncologia Medica, Avellino
  - IRCCS Istituto Tumori "Giovanni Paolo II"- U.O. Oncologia Medica, Bari
  - A.O.U. Careggi- S.C. Oncologia Medica 1, Florence
  - IRCCS A.O.U. San Martino- IST- Istituto Nazionale per la Ricerca sul Cancro- U.O.S. Tumori Polmonari, Genova
  - Ospedale Civile Livorno- U.O. Dipartimento di Oncologia Medica, Livorno
  - Ospedale Campo di Marte- U.O.C. di Oncologia Medica, Lucca
  - Istituto Europeo di Oncologia - Divisione di Oncologia Toracica, Milan
  - A.O.U. Policlinico di Modena- Oncologia Ematologia e Malattie Apparato Respiratorio, Modena
  - Istituto Nazionale per lo Studio e la Cura dei Tumori "Fondazione Giovanni Pascale"- Oncologia Medica Dipartimento Toraco-Polmonare, Napoli
  - A.O.U. "Maggiore della Carità"- Dipartimento Oncologico, Novara
  - Istituto Oncologico Veneto IRCCS- UOS Oncologia Toracica UOC. Oncologia Medica 2, Padua
  - Casa di Cura La Maddalena- U.O. Oncologia medica, Palermo
  - Azienda Ospedaliera Universitaria di Parma- Struttura Complessa di Oncologia Medica, Parma
  - Ospedale Santa Maria della Misericordia - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliero Universitaria Pisana (AOUP)- Pneumo-Oncologia - Dipartimento Cardio-Toracico, Pisa
  - Ospedale di Ravenna- Oncologia Medica, Ravenna
  - Ospedale "Infermi" Rimini- UU.OO. Oncologia ed Ematologia, Rimini
  - Osp. Civile SS. Annunziata- U.O.C di Oncologia Medica, Sassari
  - Policlinico 'G.B.Rossi' Borgo Roma - A.O.U. Integrata (Giampaolo Tortora)- Oncologia Medica, Verona

REFERENCES:
- [Derived] Chiari R, Ricciuti B, Landi L, Morelli AM, Delmonte A, Spitaleri G, Cortinovis DL, Lamberti G, Facchinetti F, Pilotto S, Verusio C, Chella A, Bonanno L, Galetta D, Cappuzzo F. ROS1-rearranged Non-small-cell Lung Cancer is Associated With a High Rate of Venous Thromboembolism: Analysis From a Phase II, Prospective, Multicenter, Two-arms Trial (METROS). Clin Lung Cancer. 2020 Jan;21(1):15-20. doi: 10.1016/j.cllc.2019.06.012. Epub 2019 Jun 18. PMID 31607443
- See also: Fondazione FoRT — http://www.fondazionefort.org/